CLINICAL TRIAL: NCT03699267
Title: Efficacy of Ultrasound-guided Transversus Abdominis Plane Block in Breast Reconstruction Surgery With Abdominal Myocutaneous Flap: an Observational Prospective Study
Brief Title: Efficacy of US-guided TAP Block in Breast Reconstruction Surgery With Abdominal Myocutaneous Flap
Status: Completed | Type: Observational
Sponsor: Instituto Portugues de Oncologia, Francisco Gentil, Porto (Other)
Responsible Party: Principal Investigator, Ana Luísa Santos Afonso, Resident of Anesthesiology, Instituto Portugues de Oncologia, Francisco Gentil, Porto
Other Study IDs: 88/561
Record Dates: First submitted 2018-10-04; First posted 2018-10-09 (Actual); Last update posted 2018-10-09 (Actual); Status verified 2018-10

CONDITIONS: Breast Reconstruction Surgery; TAP Block; Ultrasound; Analgesia; Efficacy
MeSH Terms: conditions — Agnosia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- UBR TRAM / GBA: Patients scheduled for unilateral breast reconstruction surgery with TRAM flap whose anesthetic plan adopted by the anesthetist was general balanced anesthesia
- UBR TRAM / GBA + TAP: Patients scheduled for unilateral breast reconstruction surgery with TRAM flap whose anesthetic plan adopted by the anesthetist was general balanced anesthesia combined with US-guided bilateral TAP block
  Interventions: Other: US-guided Bilateral TAP block
- M + UBR TRAM / GBA: Patients scheduled for partial/total or totalization mastectomy followed by TRAM reconstruction whose anesthetic plan adopted by the anesthetist was general balanced anesthesia
- M + UBR TRAM / GBA + TAP: Patients scheduled for partial/total or totalization mastectomy followed by TRAM reconstruction whose anesthetic plan adopted by the anesthetist was general balanced anesthesia combined with US-guided bilateral TAP block
  Interventions: Other: US-guided Bilateral TAP block

INTERVENTIONS:
Other: US-guided Bilateral TAP block
  Groups: M + UBR TRAM / GBA + TAP; UBR TRAM / GBA + TAP

SUMMARY:
Ultrasound (US)-guided transversus abdominis plane block (TAP) has demonstrated favourable results in lower abdominal surgery. Literature about its efficacy in breast reconstruction surgery with transversus rectus abdominis myocutaneous (TRAM) flap is still scarce.

In the current study investigators pretend to evaluate the efficacy of US-guided bilateral TAP block for unilateral breast reconstruction using autologous abdominal graft in women with breast cancer's history.

DETAILED DESCRIPTION:
The investigators led a prospective observational study in patients/participants scheduled to unilateral breast reconstruction surgery with TRAM flap (UBR TRAM) or partial/total or totalization mastectomy followed by TRAM reconstruction (M + UBR TRAM). Participants' anesthetic plan was general balanced anesthesia (GBA) or general balanced anesthesia combined with bilateral TAP block (GBA + TAP).

The anesthetic plan was adopted by the anaesthetist assigned to the operating room on surgery's day. Then, two groups were considered for the study: group submitted to GBA and another submitted to GBA + TAP. Anaesthetic information about intra-operative date was consulted. Investigators included patients subjected to general anesthesia with orotracheal intubation. Intravenous (IV) bolus of fentanyl were administered at anesthetic induction and according to analgesic needs. In patients whose anesthetic plan included TAP block investigators considered cases that it was performed after anesthetic induction before surgical incision. TAP block was performed according to Anesthesiology's Department. After aspiration, a volume of 20 mL ropivacaine 0.375% was administered, bilaterally. Investigators didn´t consider for the study participants whose systemic postoperative analgesic protocol wasn't that adopted by Anesthesiology Department for this kind of surgery.

It was evaluated:

* Intraoperative period: fentanyl consumption (mg/kg), antiemetic prophylaxis and anesthesia duration;
* Post-anaesthesia care unit (PACU): consumed opioids, total score and score relative to consciousness, at admission and discharge, pain assessment, at admission and discharge and nausea and vomiting incidence and stay's length
* After discharge of PACU until 4 hours after surgery's end and between 4th until 24th postoperative hour: morphine consumption, pain assessment, nausea and vomiting incidence and other complications.

ELIGIBILITY:
Inclusion Criteria:

* Patients of age superior 18 years-old;
* Patients scheduled to unilateral breast reconstruction surgery with TRAM flap or partial/total or totalization mastectomy followed by TRAM reconstruction whose anesthetic plan was GBA or GBA + TAP.

Exclusion Criteria:

* Refusal to participate in study;
* Inability to sign written informed consent;
* Body mass index superior (BMI) 40 kg/m2;
* Opioid tolerance (defined as previous consume, minimum period of 2 months, ≥ 50 mg morphine equivalents, per os);
* Substance abuse (addiction syndrome)
* Renal chronic disease with creatinine clearance < 30 mL/min/1.73m2); hepatic disease (Child-Pugh score of 1, 2 or 3);
* Patients subjected to other surgeries within the same operative time
* Patients that TAP block was not performed before surgical incision and the dose and volume of ropivacaine wasn't 20 mL, ropivacaine 0.375%
* Patients whose systemic analgesic protocol wasn't that adopted by Anesthesiology Department for this kind of surgery

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Women with age superior to 18 years-old scheduled for unilateral breast reconstruction surgery with TRAM flap or partial/total or totalization mastectomy followed by TRAM reconstruction in the study site.
Sampling Method: Non-Probability Sample
Enrollment: 107 (Actual)
Dates: Start 2015-04 (Actual); Primary Completion 2017-06 (Actual); Study Completion 2017-06 (Actual)

PRIMARY OUTCOMES:
Fentanyl consumed/administered during intraoperative time | Investigators recorded this variable for each participant since the date of start of the study until its end (since April 2015 until June 2017, 2 years and 2 months). Outcome was globally evaluated for each cohort at the end of the study (June 2017).
  Based on anaesthesia records, fentanyl administered during intraoperative time was calculated in milligrams per kilogram for each participant.
Morphine consumed/administered during post-anaesthesia care unit stay | Investigators recorded this variable for each participant since the start of the study until its end (since April 2015 until June 2017, 2 years and 2 months). Outcome was globally evaluated for each cohort at the end of the study (June 2017).
  Based on post-anaesthesia care unit records, quantity, in milligrams, of supplemental morphine administered to each participant was recorded.

SECONDARY OUTCOMES:
Morphine consumed/administered after discharge from post-anaesthesia care unit discharge until 24 hours since surgery's end | Investigators recorded this variable for each participant since the start of the study until its end (since April 2015 until June 2017, 2 years and 2 months). Outcome was globally evaluated for each cohort at the end of the study (June 2017).
  Based on records from Acute Pain Registration, it was recorded, for each participant, total morphine consumed/administered, in milligrams, since post-anaesthesia care unit's discharge until 4th postoperative hour and since 4th until 24th postoperative hour.
Pain's assessment at rest and on movement | Investigators recorded these variables for each participant since the start of the study until its end (since April 2015 until June 2017, 2 years and 2 months). Outcome was globally evaluated for each cohort at the end of the study (June 2017).
  Evaluation of pain at rest and on movement, using a qualitative scale. Investigators used qualitative pain scale adopted in the study site. Scale ranges from 0 to 4. It is defined as: 0 - no pain reported by participant; 1 - slight pain reported by participant; 2 - moderate pain reported by participant; 3 - severe pain reported by participant and 4 - excruciating pain.
  Pain assessment was recorded, based on records from post-anaesthesia care unit and Acute Pain Registration, for each participant at different moments. At admission and discharge from post-anaesthesia care unit, at 4th postoperative hour and at 24th postoperative hour.
Recovery score, at admission and discharge from post-anaesthesia care unit, according to post-anaesthesia care unit's discharge criteria | Investigators recorded these variables for each participant since the start of the study until its end (since April 2015 until June 2017, 2 years and 2 months). Outcome was globally evaluated for each cohort at the end of the study (June 2017).
  It was registered for each participant, total score at PACU's admission and discharge according to: Peripheral O2 saturation: 0 - < 85%, 1 - 85-95% and 2 - > 95%; Motor activity: 0 - inability to move, 1 - move 2 extremities; 2 - move 4 extremities; Hemodynamic: 0 - variation of medium arterial pressure (MAP) comparing to pre-anaesthetic evaluation > 40 mmHg or hear rate (HR)<40 or >50 bpm; 1 - variation of MAP comparing to pre-anaesthetic evaluation >40 mmHg or HR<50 or >120; 2 - MAP and HR similar to pre-anesthetic evaluation; Temperature: 0 - body temperature (T)<35ºC; 1 - T 35-35.5ºC; 2 - T 35.5-36ºC; Breathing: 0 - no spontaneous breathing; 1 - dyspnea/respiratory rate (RR) <10 or >20; 2 - eupnea; Consciousness: 0 - nor responding to stimuli; 1 - responding to simple questions; 2 - awake and alert; Nausea/Vomiting: 0 - vomiting; 1 - nausea; 2 - no nausea or vomiting; Pain: 0 - intolerable; 1 - intense; 2 - mild; 3 - no pain. Total score was calculated by summing each score.
Nausea and vomiting incidence | Investigators recorded these variables for each participant since the start of the study until its end (since April 2015 until June 2017, 2 years and 2 months). Outcome was globally evaluated for each cohort at the end of the study (June 2017).
  Based on post-anaesthesia care unit and ward records, it was registered any episodes of nausea or vomiting for each participant until 24th postoperative hour.

CONTACTS AND LOCATIONS:
Overall Officials: Ana Afonso, Principal Investigator — IPO-Porto, E.P.E.